CLINICAL TRIAL: NCT05375422
Title: Effects of the Strengthening and Stretching Protocol for Rheumatoid Arthritis in the Hands (SARAH) on Hand Function in Women With Rheumatoid Arthritis
Brief Title: Effects of SARAH Protocol in Women With Rheumatoid Arthritis
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Federal University of Espirito Santo (Other)
Responsible Party: Principal Investigator, Samira Tatiyama Miyamoto, PhD, Professor, Federal University of Espirito Santo
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: FUEspiritoSanto03
Record Dates: First submitted 2022-05-11; First posted 2022-05-16 (Actual); Last update posted 2022-05-16 (Actual); Status verified 2022-05

CONDITIONS: Rheumatoid Arthritis
Keywords: exercise; hand; physical therapy
MeSH Terms: conditions — Arthritis, Rheumatoid; Motor Activity | interventions — Early Intervention, Educational

STUDY DESIGN:
Who Masked: Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- SARAH group (Experimental): The SARAH group will receive an exercise book containing 7 mobility exercises and 4 strength exercises that are performed using elastic materials that provide progressive degrees of resistance to movement. Patients will be guided in person by a trained professional, so that they are carried out without their presence, in the home environment, daily and monitored at periodically scheduled meetings. A total of 4 face-to-face meetings will be held during the 3-month follow-up. The SARAH group and the control group will receive information related to joint protection, use of splints, assistive devices and other general advice, as needed, will receive some booklets to reinforce the guidelines. The program will last 12 weeks, with 4 face-to-face meetings lasting 40 minutes and monitored in periodically scheduled meetings.
  Interventions: Other: SARAH; Other: Educational intervention
- Control group (Active Comparator): Control group will receive information related to joint protection, use of splints, assistive devices and other general advice, as needed, will receive some booklets to reinforce the guidelines.
  After 12 weeks, the control group will also be invited to perform the SARAH protocol exercises.
  Interventions: Other: Educational intervention

INTERVENTIONS:
Other: SARAH — Set of exercises with components of muscle strengthening, range of motion gain and home exercises.
  Arms: SARAH group
Other: Educational intervention — Information related to joint protection, use of splints, assistive devices and other general advice, as needed.

SUMMARY:
The aim of this randomized controlled trial is to analyze the effect of the SARAH protocol, which is a set of exercises with components of muscle strengthening, range of motion gain and home exercises, combined with an educational intervention, on hand function in women with rheumatoid arthritis (RA).

DETAILED DESCRIPTION:
The volunteers will be randomized between groups: control group (n=30), which will receive usual guidelines and the SARAH group (n=30), which will perform the SARAH protocol exercises (brazilian portuguese version) along with the usual guidelines. To participate in the research, patients must be diagnosed with RA using disease-modifying antirheumatic medication for at least 3 months, and age equal to or older to 18 years. Participants with incomplete elementary school and score <24 on the Mini-Mental State Examination Questionnaire (MMSE) will be excluded from the study. The participants will be evaluated before and after the intervention regarding the variables: hand function (Michigan Hand Outcomes Questionnaire), pain (Brief Pain Inventory), handgrip strength (Jamar® manual dynamometer), quality of life (Euro Quality of Life Instrument-5D), functional capacity (Health Assessment Questionnaire), RA disease activity (DAS28). The SARAH group will receive an exercise book containing 7 mobility exercises and 4 strength exercises that are performed using elastic materials that provide progressive degrees of resistance to movement. Patients will be guided in person by a trained professional, so that they are carried out without their presence, in the home environment, daily and monitored at periodically scheduled meetings. A total of 4 face-to-face meetings will be held during the 3-month follow-up. The SARAH group and the control group will receive information related to joint protection, use of splints, assistive devices and other general advice, as needed, will receive some booklets to reinforce the guidelines. The program will last 12 weeks, with 4 face-to-face meetings lasting 40 minutes and monitored in periodically scheduled meetings.

ELIGIBILITY:
Inclusion Criteria:

* patients must be diagnosed with RA
* using disease-modifying antirheumatic medication for at least 3 months
* over 18 years old

Exclusion Criteria:

* incomplete elementary school and score <24 on the Mini-Mental State Examination Questionnaire (MMSE)
* diagnosis of another associated autoimmune disease
* having undergone previous surgical procedures on the hands
* having suffered a fracture in the joints of the upper limbs in the last six months
* being a patient on the waiting list for orthopedic surgery of the upper limb
* being pregnant.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — women over 18 years old
Enrollment: 60 (Estimated)
Dates: Start 2022-02-07 (Actual); Primary Completion 2022-05-07 (Actual); Study Completion 2024-02-07 (Estimated)

PRIMARY OUTCOMES:
Hand function | 3 months
  Michigan Hand Outcomes Questionnaire. A total of 37 items assess six domains: general hand function, activities of daily living, work performance, pain, aesthetics, and patient satisfaction with hand function. The participant must score each item using Likert-type scales ranging from 1 to 5.

SECONDARY OUTCOMES:
Pain inventory | 3 months
  Brief Pain Inventory. It classifies pain as mild when scored from 1 to 4, moderate when scored from 5 to 7, and severe when the participant selects values from 8 to 10 points.
Hand grip strength | 3 months
  Hand dynamometer. The participant should press the dynamometer with maximum force for 3 seconds and rest for 60 seconds. All values must be recorded for later calculation of the average of three attempts.
Healthy related quality of life | 3 months
  Euro Quality of Life Instrument-5D (EQ-5D). The questionnaire consists of questions about health and disease states, such as: mobility, personal care, usual activities, pain/discomfort, anxiety/depression, and each of these has three associated levels of severity, corresponding to no problems (level 1). ), some problems (level 2) and extreme problems (level 3) experienced or felt by the individual.
Functional capacity | 3 months
  Health Assesment Questionnaire (HAQ). Eight categories with scores from 0 (no problem) to 3 (unable to do) per category. The score for each category appears at the highest number of any of its items, and the final HAQ score is the average of the scores for the eight categories.
Disease activity | 3 months
  Disease Activity Score (DAS-28). The DAS-28 score can be interpreted on a categorical scale: it is indicative of disease remission values <2.6, light activity when it has a result between 2.6 and 3.2, moderate activity when values >3.2 to 5, 1 and high disease activity when the result is greater than 5.1.

CONTACTS AND LOCATIONS:
Locations (1):
- Samira Tatiyama Miyamoto, PhD, Vitória, Espírito Santo, Brazil

IPD SHARING:
Plan to Share IPD: No